CLINICAL TRIAL: NCT00890084
Title: RESPECT: Observational, Prospective, Open-label, Multi-center Study Evaluating the Antihypertensive Effect of Treatment With Telmisartan (Alone or in Fixed Combination With HCTZ) in General Practitioner and Specialist Practice in Hypertensive Patients With High and Very High Cardiovascular Risk According to the ESH/ESC Guidelines 2007 Who Are Uncontrolled Under Current Treatment.
Brief Title: Telmisartan Tab Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.581
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan, hydrochlorothiazide drug combination

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group1
  Interventions: Drug: Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)

INTERVENTIONS:
Drug: Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ) — Telmisartan 40mg or 80mg +/- HCTZ 12.5mg or 25mg

SUMMARY:
To assess the efficacy of telmisartan in hypertensive patients with high cardiovascular risk

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion criteria:

Hypertensive patients with BP. 140/90mmHgand high and very high cardiovascular risk according to the ESH/ESC Guidelines 2007 and in whom the prescriber has taken the decision to start treatment with telmisartan 40 or 80 mg, with or without HCTZ 12.5 mg or 25 mg, in the usual way and in line with the SmPC and reimbursement criteria

Exclusion criteria:

Contra-indications as in the Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 2913 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 1st 2009 to January 1st 2010 recruited in 90.5% General Practitioners (GP's) and 9.5% Specialists (Sp's)
Pre-assignment Details: 45 patients excluded for inclusion/exclusion criteria
Period: Overall Study
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Started | 2913
Completed | 2771
Not Completed | 142
Not completed — Adverse Event | 16
Not completed — Lost to Follow-up | 126

BASELINE CHARACTERISTICS:
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 2913
Age, Customized [Mean (Standard Deviation); unit: years] | 64.4 (12.6)
Sex/Gender, Customized [Number; unit: percentage of participants]
  Female | 48.8
  Male | 51.2
Systolic and diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic Blood Pressure | 156.1 (12.9)
  Diastolic Blood Pressure | 91.9 (8.64)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Blood Pressure < 140/90 mm Hg
Description: % of high risk patients with Blood Pressure < 140/90 mm Hg
Time Frame: 12 weeks
Population: Intention-to-Treat (ITT)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 2771
Percentage of participants | 69.6 [67.9 to 71.3]

2. Secondary Outcome: Percentage of Patients With Blood Pressure < 130/80 mm Hg
Time Frame: 12 weeks
Population: Intention to Treat (ITT)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 2771
Percentage of participants | 13.2 [12.0 to 14.5]

3. Secondary Outcome: Absolute Blood Pressure Decrease
Description: systolic blood pressure
Time Frame: baseline and 12 weeks
Population: Intention to treat (ITT)
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 2771
mm Hg | 23.2 [22.7 to 23.7]

4. Secondary Outcome: BP Response Rate (Drop of Systolic BP of 10mmHg or More)
Description: BP response rate (drop of systolic BP of ≥ 10mmHg) after approximately 12 weeks of treatment with telmisartan (alone or in fixed combination with HCTZ)
Time Frame: 12 weeks
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 2771
Percentage of patients | 91.85 [90.8 to 92.6]

5. Secondary Outcome: Treatment Patterns
Description: Treatment patterns observed at the end of the study as Micardis monotherapy, Micardis Plus 12.5 and Micardis Plus 25 (with or without changes in concomitant antihypertensive medications).
Time Frame: 12 weeks
Population: ITT Population
Measure: Number; unit: Percentage of patients
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 2771
Percentage of patients
  Telmisartan 40mg | 4.7
  Telmisartan 80mg | 49.4
  Telmisartan 40/12,5mg | 3.3
  Telmisartan 80/12,5mg | 29.7
  Telmisartan 80/25mg | 12.6

6. Secondary Outcome: Change in Concomitant Antihypertensive Drugs Given at Study Entry
Description: Percentage of patients who had a change in concomitant antihypertensive drugs prescribed at initiation and after 12 weeks. The antihypertensive drugs were changed (which is stopped, titration of dose and started) or not.
Time Frame: baseline and 12 weeks
Population: Intention to treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 2771
percentage of patients | 13.6 [12.3 to 14.9]

7. Secondary Outcome: Percentage of Patients in Whom the Prescriber Decide to Further Lower the Blood Pressure to < 130/80 mm Hg
Time Frame: 12 weeks
Population: Intention to treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 2771
percentage of patients | 11.7 [10.5 to 12.9]

8. Secondary Outcome: Percentage of Prescribers Who Adhered to European Society of Hypertension/European Society of Cardiology (ESH/ESC) Guidelines 2007
Description: Blood pressure should be reduced to at least below 140/90 mm Hg (systolic/diastolic),and to lower values, if tolerated, in all hypertensive patients. Target blood pressure should be lower than 130/80 mmHg in diabetics and in high or very high risk patients
Time Frame: 12 weeks
Population: all investigators participating in the trial
Measure: Number (95% Confidence Interval); unit: percentage of prescribers
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Number analyzed (Participants) | 432
percentage of prescribers | 47.7 [43 to 52.4]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: solicited reporting
Arm/Group | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ)
Serious Adverse Events (participants affected / at risk) | 3/2771
Other Adverse Events (participants affected / at risk) | 0/2771
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan or Telmisartan + Hydrochlorothiazide (HCTZ) (N=2771)
Umbilical hernia (Gastrointestinal disorders) | 1
Alcohol detoxification (Surgical and medical procedures) | 1
cerebral hemorrhage, fatal (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.